CLINICAL TRIAL: NCT05247684
Title: Phase II Clinical Study of AK112, an Anti-PD-1 and VEGF Bispecific Antibody, Alone or in Combination With Chemotherapy for the Neoadjuvant/Adjuvant Treatment of Resectable Non-small Cell Lung Cancer
Brief Title: AK112 Neoadjuvant/Adjuvant Treatment for Resectable NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-205
Record Dates: First submitted 2022-01-19; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Resectable Non-small Cell Lung Cancer
MeSH Terms: interventions — Carboplatin; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm 1(AK112) (Experimental): Neoadjuvant therapy was 3-4 cycles of AK112(Q3W), followed by surgery ,followed by adjuvant therapy for 16 cycles of AK112(Q3W)
  Interventions: Drug: AK112
- arm 2(AK112+Carboplatin/cisplatin + paclitaxel) (Experimental): Neoadjuvant therapy was 3-4 cycles of AK112 plus Carboplatin/cisplatin + paclitaxel(Q3W), followed by surgery ,followed by adjuvant therapy for 16 cycles of AK112(Q3W)
  Interventions: Drug: AK112; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: AK112 — IV infusion
Drug: Carboplatin — IV infusion
  Arms: arm 2(AK112+Carboplatin/cisplatin + paclitaxel)
Drug: Cisplatin — IV infusion
  Arms: arm 2(AK112+Carboplatin/cisplatin + paclitaxel)
Drug: Paclitaxel — IV infusion
  Arms: arm 2(AK112+Carboplatin/cisplatin + paclitaxel)

SUMMARY:
AK112, alone or in combination with chemotherapy for the neoadjuvant/adjuvant treatment of resectable NSCLC

DETAILED DESCRIPTION:
Phase II clinical study of AK112, an anti-PD-1 and VEGF bispecific antibody, alone or in combination with chemotherapy for the neoadjuvant/adjuvant treatment of resectable non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1、18 to 75 years old

2、Be able and willing to provide written informed consent and to comply with all requirements of study participation

3、Histologically confirmed resectable stage II-IIIB NSCLC

4、Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

5、Has adequate organ function

6、All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

1. Is currently participating in a study of an investigational agent or using an investigational device
2. Has an active autoimmune disease that has required systemic treatment in the past 2 years
3. Has an active infection requiring systemic therapy
4. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
5. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
6. Has received a live virus vaccine within 30 days prior to first dose of study treatment
7. Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2023-08-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE) | Up to approximately 2 years
  Summary of AE incidence; summary after grading of AE according to NCI CTCAE version 5.0
rate of surgical delays | Up to approximately 2 years
  Proportion of subjects exceeding the maximum surgical time window
abnormal laboratory findings of clinical significance | Up to approximately 2 years
  Proportion of subjects with abnormal and clinically significant results including routine blood tests, blood biochemical tests, coagulation tests, thyroid function tests, routine urine tests, pregnancy tests, etc.
MPR | Up to approximately 2 years
  Proportion of subjects with ≤10% residual live tumor cells in resected primary tumor foci and lymph nodes

SECONDARY OUTCOMES:
R0 resection rate | Up to approximately 2 years
  Proportion of subjects with pathologically complete resection of primary tumors
Tumor descending stage rate | Up to approximately 2 years
  Proportion of subjects with the most recent tumor staging prior to surgery (using TNM staging version 8) who were down-staged relative to baseline
pCR | Up to approximately 2 years
  Proportion of subjects with no residual tumor in the resected tumor primary and lymph nodes
OS | Up to approximately 2 years
  Time from first dose until death from any cause
EFS | Up to approximately 2 years
  Time from first dose to the occurrence of any of the following events, whichever occurs first: disease progression, local recurrence or distant metastasis or death from any cause, as assessed according to RECIST v1.1.
ORR | Up to approximately 2 years
  ORR is the proportion of subjects with CR or PR,based on recist v1.1